CLINICAL TRIAL: NCT07390305
Title: Study on the Correlation Between Skin Aging in Exposed / Non Exposed Areas and Menopausal Symptoms, Emotions, and Sleep in Menopausal Women
Brief Title: Multidimensional Correlation Study on Skin Aging in Menopausal Women
Status: Completed | Type: Observational
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Other Study IDs: W25006001
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Skin Aging; Reproductive Aging; Menopause; Genetic Factors
Keywords: Skin Aging; Reproductive Aging; Menopause; Exposed/Non-Exposed Skin Sites; Hormonal Fluctuations; Genetic Factors; Mother-Daughter Pairs; Longitudinal Tracking; Skin Biophysical Properties

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early Perimenopausal Group
- Late Perimenopausal Group
- Postmenopausal Group
- Young Control Group

SUMMARY:
Primary Objective:

This study primarily aims to compare skin aging characteristics between women at different stages of reproductive aging in both sun-exposed and non-exposed areas, based on skin indicators collected during a single laboratory visit. Furthermore, through a 30-day at-home tracking period (for the late-stage and postmenopausal groups) or one menstrual cycle (for the early-stage and young group), we seek to analyze the temporal dynamics of changes in skin condition, mood, sleep quality, and menopausal hot flashes.

Secondary Objective:

The secondary objective is to examine differences in skin conditions across life stages by recruiting mother-daughter pairs (where the young group consists of the biological daughters of the late-stage and postmenopausal groups). The core focus is to leverage shared genetic backgrounds to explore how skin characteristics, particularly in different body areas, may change over time or in response to hormonal fluctuations. By comparing these characteristics across age groups, this study seeks to identify key variation patterns and their contributing factors, thereby laying the groundwork for further mechanistic investigations and practical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must possess basic Chinese literacy skills (reading comprehension and expression) to complete questionnaires independently.
2. Voluntary participation and signed informed consent.
3. Willingness to comply with all study requirements and assessments.
4. Early Perimenopausal Group：

   1. Healthy women aged 45-50 (±3) years.
   2. STRAW Stage -2 / Early Perimenopause: Experiencing a persistent change in menstrual cycle length of >7 days from their normal cycle, but with no occurrence of 60 or more days of amenorrhea (i.e., still having menstrual periods).
5. Late Perimenopausal Group：

   1. Healthy women aged 50-55 (±3) years.
   2. STRAW Stage -1 / Late Perimenopause: Experiencing ≥2 consecutive cycles with a length of ≥60 days, or the presence of ≥60 days of amenorrhea.

      6) Postmenopausal Group：

   <!-- -->

   1. Healthy women aged 55-60 (±3) years.
   2. STRAW Stage +1 / Postmenopause: Last menstrual period occurred at least 12 months prior.

7）Young Control Group：

1. Healthy women aged 18-25 (±3) years.
2. Biological daughters of participants in either the Late Perimenopausal Group or the Postmenopausal Group.
3. Regular menstrual cycle, with a cycle length ranging between 25-35 days. Exclusion Criteria

   1. Presence of open wounds, clearly visible scars, acne marks, or other significant skin imperfections at the measurement sites.
   2. History of skin diseases affecting the evaluation of the study areas (e.g., psoriasis, atopic dermatitis, skin cancer).
   3. Women who are currently pregnant or breastfeeding.
   4. Use of systemic estrogen or progesterone hormone replacement therapy within the past 6 months.
   5. Presence of acute or severe chronic diseases currently under treatment.
   6. Any known condition that significantly impairs cognitive or behavioral abilities.
   7. Considered by the investigator or qualified professional to have other medical or specific reasons that may interfere with the evaluation of study results.
   8. Early Perimenopausal Group & Late Perimenopausal Group & Postmenopausal Group:

a) Current use of systemic hormone replacement therapy (HRT). b) Topical application of anti-aging products (e.g., retinoids, alpha/beta hydroxy acids) on the measurement areas within the past 3 months.

c) History of breast cancer or oophorectomy. 9） Young Control Group:

1. Currently planning for pregnancy, pregnant, or lactating.
2. Diagnosis of Polycystic Ovary Syndrome (PCOS).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study enrolled adult women categorized into four distinct groups based on their reproductive aging stage according to the STRAW+10 staging system: a Young Control Group (aged 18-25, biological daughters of participants in the older groups, with regular menstrual cycles), an Early Perimenopausal Group (aged 45-50, with a persistent change in menstrual cycle length >7 days), a Late Perimenopausal Group (aged 50-55, experiencing ≥2 consecutive cycles of ≥60 days or amenorrhea of ≥60 days), and a Postmenopausal Group (aged 55-60, with the last menstrual period occurring at least 12 months prior). All participants were recruited as mother-daughter pairs, where the young control group consisted of the biological daughters of participants in the late perimenopausal and postmenopausal groups .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment | The assessment is performed as a single evaluation at the T1 (baseline) laboratory visit .
  This assessment involves a clinical evaluation of skin aging degree performed by dermatologists at the T1 time point. The evaluation is conducted according to the skin aging scales outlined in the "Human Skin Aging Evaluation Standard" . It targets both exposed areas (face, dorsum of hands) and non-exposed areas (inner side of the upper arm, outer upper hip region) to differentiate between intrinsic and extrinsic aging factors. Specific skin lesions, such as epidermal/vascular proliferations, are assessed as separate individual items.
Skin Wrinkle and Smoothness Assessment | The assessment is conducted as a single measurement at the T1 (baseline) time point .
  This assessment quantitatively evaluates skin surface topography using a dedicated imaging system. The instrument captures high-resolution grayscale images of the skin's surface. The built-in Skin Evaluation Living Skin (SELS) software then analyzes the image to extract objective numerical values for key parameters. The primary indicators measured are: SEw (Surface Evaluation of Wrinkles), where a higher value indicates more pronounced wrinkles; and SEsm (Surface Evaluation of Smoothness), where a lower value indicates smoother skin.
Skin Color Measurement with Colorimeter | The measurement is performed as a single assessment at the T1 (baseline) laboratory visit.
  This assessment quantitatively measures skin color using the Colorimeter probe. The instrument emits white LED light from a ring-shaped configuration to ensure even illumination of the skin surface. The light scatters upon contact, with some penetrating the skin and some being reflected. The probe captures the reflected light, and the raw data is corrected via a specialized color matrix to approximate standard values. The skin color is expressed in XYZ tristimulus values and converted into the standardized CIE Lab* color space parameters. The L* value represents lightness (brightness) on a black-white axis. The a* value indicates the position on the red-green axis (often interpreted as erythema or red pigment), and the b* value indicates the position on the blue-yellow axis (often associated with yellow pigment). Additionally, the Individual Typology Angle (ITA°) value is automatically calculated, where a higher ITA° value indicates lighter skin.
Skin Elasticity Measurement with Cutometer® MPA580 | The measurement is performed as a single assessment at the T1 (baseline) laboratory visit .
  The Cutometer® MPA580 assesses skin mechanical properties based on the suction and stretch principle. It applies a controlled negative pressure to the skin, drawing it into the probe aperture. The depth of skin deformation is measured optically by the ratio of light emitted to light received within the probe. Key parameters extracted for this study include R2 (Gross Elasticity) and F4 (Firmness). The R2 value, representing the ratio of total retraction to total deformation, approaches 1 for highly elastic skin. The F4 value corresponds to the skin's firmness or resistance to the suction force; a lower F4 value indicates firmer, more resistant skin .
Skin Ultrasound Diagnostic System Ultrascan UC22 | The measurement is performed as a single assessment at the T1 (baseline) laboratory visit.
  The Ultrascan UC22 is a high-frequency ultrasound imaging system used for non-invasive assessment of skin microstructure. It operates by emitting a 22 MHz ultrasound signal into the skin; the echoes reflected from internal skin structures are captured and digitally processed to generate high-resolution, cross-sectional images. This allows for the in vivo measurement of key parameters related to skin aging, primarily skin thickness and skin density (which correlates with collagen density and tissue structure). This tool is particularly valuable for objectively evaluating intrinsic skin aging and the efficacy of cosmetic interventions in research settings.
Skin Moisture Loss Meter Vapometer | The measurement is performed as a single assessment at the T1 (baseline) laboratory visit .
  he Vapometer is a portable device designed to measure Transepidermal Water Loss (TEWL), a key indicator of the skin barrier's functional integrity. Its operation is based on the closed-chamber principle. The core of the instrument is a highly sensitive humidity sensor located within a cylindrical measurement chamber. During measurement, this chamber is sealed against the skin surface, creating a microenvironment protected from ambient air currents. The sensor monitors the increase in relative humidity (RH) inside the chamber caused by the evaporation of water from the skin. The TEWL value, expressed in grams per square meter per hour (g/m²h), is automatically calculated from this rate of humidity increase . This method is particularly suitable for detecting changes in skin water loss and is widely used in dermatological research and cosmetic efficacy evaluations.
Skin Hemoglobin Measurement with Mexameter® MX18 | The assessment is performed as a single measurement at the T1 (baseline) laboratory visit .
  The Mexameter® MX18 is a specialized probe that quantitatively assesses skin color by measuring the two primary chromophores: melanin and hemoglobin. It operates on the principle of light absorption and reflection.
Intelligent Skin Analyzer Skinmeter | The measurement is performed at three designated time points during the study: T1( Day1),T2(Day 15), and T3(Day 30).
  The Skinmeter is a portable device designed for the non-invasive assessment of key skin physiological parameters. For the purpose of this study, the primary focus of the measurement is on the skin hydration (moisture) parameter.
Skin Sebum Measurement with Sebum-Test Paper | The measurement is performed at three designated time points during the study: T1( Day1),T2(Day 15), and T3(Day 30).
  This method quantitatively assesses skin sebum (oil) content using a specialized oil-absorbent test paper and subsequent image analysis.
Sleep Duration Recording | Sleep data is collected continuously throughout the entire tracking period of the study.Day1 to Day 30.
  This component utilizes the smart band monitoring algorithm to objectively record participants' sleep patterns. The algorithm employs a multi-modal approach, integrating data from accelerometers (to monitor body movement) and photoplethysmography (PPG) sensors (to monitor heart rate and heart rate variability) . By analyzing the correlation between physiological signals such as body movement, heart rate, and their variability with sleep states, it constructs a fusion algorithm model to accurately identify sleep stages and calculate total sleep duration . This non-invasive method allows for convenient, at-home sleep monitoring over extended periods.

SECONDARY OUTCOMES:
BMI | BMI is measured during the baseline laboratory visit.
  Body Mass Index (BMI) is a widely used international standard for assessing body weight and health status. It is a numerical value calculated from an individual's weight and height.
Pittsburgh Sleep Quality Index (PSQI) | The PSQI questionnaire will be administered at three designated time points during the study: Day1, Day15, and Day30. At each assessment, participants will be asked to recall and report on their sleep quality and disturbances over the past 1 week .
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire widely used to assess subjective sleep quality over a specified period.
Generalized Anxiety Disorder-7 (GAD-7) | he questionnaire is administered at three designated time points during the study: T1(Day1), T2(Day15), and T3(Day30). At each assessment, participants are asked to recall and report on their experiences over the past two weeks .
  The Generalized Anxiety Disorder-7 (GAD-7) is a self-report questionnaire utilized for screening and assessing the severity of generalized anxiety disorder. As a component of the Patient Health Questionnaire (PHQ) series, it consists of 7 items that inquire about the frequency of core anxiety symptoms-such as feeling nervous, anxious, or on edge, and being unable to control worrying-over a specified period. Respondents rate each item on a 4-point scale. The total score (ranging from 0 to 21) helps categorize anxiety severity, facilitating initial assessment and monitoring of symptoms.
Patient Health Questionnaire-8 Items (PHQ-8) | The questionnaire is administered at three specific time points during the study: T1 (Day1), T2(Day15), and T3(Day30). At each assessment, participants are asked to report on their experiences over the past two weeks .
  The Patient Health Questionnaire-8 (PHQ-8) is a standardized self-report instrument widely used to screen for and measure the severity of depressive symptoms . It consists of 8 items that correspond to the diagnostic criteria for depressive disorders. Respondents rate the frequency of each symptom over a specified recall period on a 4-point scale (0 to 3). The total score, ranging from 0 to 24, helps categorize depressive severity, from none to severe . It is a reliable and valid tool for use in both clinical and research settings.
Assessment of Hot Flash Frequency and Impact on Daily Life | This questionnaire is to be completed daily throughout the testing period. Participants are asked to recall and report on their hot flash experiences over the past 24 hours.From Day1 to Day30.
  This questionnaire is designed to assess the frequency and subjective impact of hot flashes (also known as vasomotor symptoms) on an individual's daily life. The instrument draws on core concepts from established tools, including the Kupperman Menopausal Index (KMI) and the Hot Flush Rating Scale (HFRS). It evaluates two primary dimensions: 1) the frequency of hot flash episodes over a specified period, and 2) the degree of interference these symptoms cause to various aspects of daily living, such as work, mood, sleep, and social activities. The aim is to provide a quantitative and qualitative measure of the burden of hot flashes
Ultraviolet (UV) Exposure Questionnaire | The questionnaire assesses UV exposure behaviors and sun protection habits over the past 1 month and is administered at the T1 (baseline) laboratory visit.
  This component quantitatively evaluates participants' real-life exposure to ultraviolet (UV) radiation and their photoprotection practices over a specified period. It encompasses key dimensions such as: 1. Sun Protection Behaviors: Frequency of use and types of physical protection (e.g., wide-brimmed hats, long-sleeved clothing) and sunscreen (including Sun Protection Factor, or SPF). 2. Outdoor Activity Patterns: Time spent outdoors for both occupational and recreational activities. The aim is to estimate individual UV exposure dose and identify potential risk factors for skin damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No